CLINICAL TRIAL: NCT05446675
Title: Single-Center Observational Study With Comparison of Endoscopic Extended-View Totally Extraperitoneal Prosthesis (eTEP) Versus Open Rives-Stoppa Repair as a Treatment of Midline Abdominal Wall Hernias With Rectus Diastasis
Brief Title: Endoscopic eTEP Versus Open Rives-Stoppa
Status: Completed | Type: Observational
Sponsor: AZ Alma (Other)
Responsible Party: Sponsor
Other Study IDs: EC/EH/220608-SK
Record Dates: First submitted 2022-06-27; First posted 2022-07-07 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Hernia, Ventral; Rectus Diastasis
Keywords: eTEP; Retromuscular; Minimally invasive; Endoscopic; Hernia; Rectus diastasis; Rives-Stoppa
MeSH Terms: conditions — Hernia, Ventral; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- eTEP: First 30 participants who meet the inclusion criteria and do not exhibit any of the exclusion criteria will be investigated. The option for endoscopic eTEP repair, if feasible, is given preoperatively as a standard for the treatment of symptomatic midline abdominal wall hernias with concomitant rectus abdominis diastasis as an alternative to open Rives-Stoppa mesh repair. The modality of operative treatment is made in cooperation with the participant.
  Interventions: Procedure: Endoscopic eTEP
- Rives-Stoppa, control: Thirty participants will be selected out of all patients who underwent an open Rives-Stoppa (midline repair with sublay mesh) in the investigators' center and who do not meet any of the exclusion criteria. Participant selection will consist of matching to participants in group 1 according to gender and age (e.g. a male participant in group 1 will be matched to a male participant (group 2) out of the investigators' records who underwent an open Rives-Stoppa repair and whose age most closely resembles the age of the matched participant in group 1).
  Interventions: Procedure: Open Rives-Stoppa

INTERVENTIONS:
Procedure: Endoscopic eTEP — Endoscopic extended view totally extraperitoneal prosthesis repair.
  Groups: eTEP
Procedure: Open Rives-Stoppa — Open Rives-Stoppa repair with retromuscular mesh placement.
  Groups: Rives-Stoppa, control

SUMMARY:
Observational cohort study (partially retrospective, partially prospective) comparing the endoscopic extended totally extraperitoneal prosthesis (eTEP) repair for midline abdominal hernias to open Rives-Stoppa repair (control).

DETAILED DESCRIPTION:
See included study protocol. Included patients will be registered to the European Hernia Society (EHS) registry.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (eTEP):

* Participants who underwent an eTEP procedure in the investigators' center
* Preoperative existence of one or more midline abdominal wall hernias
* Preoperative existence of rectus abdominis diastasis

Group 2 (Rives-Stoppa, control group):

- Participants who underwent an open Rives-Stoppa (midline repair with sublay mesh) in the investigators' center

Exclusion Criteria:

Group 1 (eTEP):

* Preoperative absence of midline abdominal wall hernias
* Preoperative absence of rectus abdominis diastasis
* Intraoperative performance of transverse abdominis release (TAR)
* Intraoperative inguinal hernia repair

Group 2 (Rives-Stoppa, control group):

* Intraoperative performance of transverse abdominis release (TAR)
* Intraoperative performance of anterior component separation
* Intraoperative inguinal hernia repair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who underwent repair for their midline abdominal wall hernias alongside rectus abdominis diastasis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | From the date of operation until the date of discharge from the hospital, assessed up to 30 days.
  Time (days) spent within the hospital
Postoperative pain management | From the end of surgery (moment of the end of operation) until the date of discharge from the hospital, assessed up to 30 days.
  Modality (type, generic name), duration (days), dosage (grams or milligrams) and frequency (times per day) of analgesics administration

SECONDARY OUTCOMES:
Intraoperative complications | During surgery
  Adverse event occurrence
Postoperative complications | After discharge until 30 days postoperative
  Adverse event occurrence by readmission

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kinet, MD, Principal Investigator — AZ Alma
Locations (1):
- AZ Alma, Eeklo, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be sent to journal at time of application for publication after completion.
  IPD will be shared via the online EHS registry with contents adhering to their format. Accessible to all EHS members for all types of analyses.
Supporting Information: Study Protocol, ICF
Time Frame: At completion of the study.
Access Criteria: EHS-membership.
URL: https://ehs-hernia-registry.com/

REFERENCES:
- [Derived] Kinet S, Maes H, Van Cleven S, Brusselaers N, Kuppens EFP. Endoscopic enhanced-view totally extraperitoneal prosthetic (eTEP) versus open Rives-Stoppa repair as a treatment of midline abdominal wall hernias with rectus diastasis: comparison of postoperative pain and length of hospital stay in a single-centre surgical cohort. Updates Surg. 2024 Dec;76(8):2923-2931. doi: 10.1007/s13304-024-01905-4. Epub 2024 Jun 23. PMID 38909352
- Available data/document: Individual Participant Data Set: EC/EH/220608-SK — https://ehs-hernia-registry.com

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-12-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT05446675/Prot_ICF_001.pdf